CLINICAL TRIAL: NCT02559141
Title: Non-invasive Early Goal Directed Therapy in Colorectal Surgery: a Feasibility Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Schleswig-Holstein (Other)
Responsible Party: Principal Investigator, Ole Broch, MD, Priv.-Doz. Dr. med. Ole Broch, University Hospital Schleswig-Holstein
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AZ B260/11
Record Dates: First submitted 2015-09-23; First posted 2015-09-24 (Estimated); Last update posted 2015-10-29 (Estimated); Status verified 2015-10

CONDITIONS: Perioperative/Postoperative Complications; C.Surgical Procedure; Digestive System
Keywords: haemodynamic optimization; cardiac index; non-invasive; pulse pressure variation
MeSH Terms: conditions — Postoperative Complications | interventions — Dobutamine; Norepinephrine; Crystalloid Solutions; Colloids

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Study group (SG) (Other): Before induction of anaesthesia:
  * Arterial line
  * Nexfin Monitoring System
  * Measurement of cardiac index (CI), pulse pressure variation (PPV) and mean arterial pressure (MAP)
  * Baseline blood samples. Induction of anaesthesia
  Study Group:
  * PPV ≤10%, 500 ml of crystalloids/colloids as long as CI was ≥2.5 l/min/m²
  * Maintenance of CI ≥2.5 l/min/m² and MAP ≥65 mmHg by using dobutamine (10 µg/kg/min) and norepinephrine (0.03 µg/kg/min).
  Interventions: Drug: Dobutamine
- Control group (CG) (No Intervention): * MAP ≥65 mmHg
  * CVP ≤12 mmHg
  * Haemoglobin level ≥8 g/dl.
  * Maintenance of MAP ≥65 mmHg by using crystalloids/colloids, bolus injection of theodrenaline/cafedrine or continuous infusion of norepinephrine (0.03 µg/kg/min) according to clinical evaluation.

INTERVENTIONS:
Drug: Dobutamine — If PPV ≤10%, volume substitution of 500 ml of crystalloids and/or colloids as long as CI was ≥2.5 l/min/m². Maintenance of CI ≥2.5 l/min/m² and MAP ≥65 mmHg was achieved by using dobutamine (10 µg/kg/min) and norepinephrine (0.03 µg/kg/min).
  Other Names: Norepinephrine; crystalloids/colloids
  Arms: Study group (SG)

SUMMARY:
The Nexfin monitoring system offers a complete non-invasive approach to a continuously estimation of blood pressure, CI and PPV by means of finger-cuff based pulse contour analysis. Several clinical investigations have proven reliability and interchangeability of the Nexfin technology yielding acceptable results especially regarding the trending abilities. At present there is no evidence available, whether a early goal directed hemodynamic optimization protocol based on a completely non-invasive monitoring technology is able to reduce postoperative complication. Therefore, the aim of this single-center study is to compare the clinical outcome and postoperative complications of patients undergoing major colorectal surgery treated with standard of care or with a GDT protocol based on the Nexfin technology.

DETAILED DESCRIPTION:
The Nexfin™ monitoring system is able to provide continuous beat-to-beat stroke volume index (SVI), stroke volume variation (SVV), pulse pressure variation (PPV), cardiac index (CI) and arterial pressure by using an inflatable finger cuff. This system consists of a frequency dependent transfer function for calculation of brachial artery pressure from the finger artery pressure.

Major surgery bares the risk of concealed hypoperfusion and therefore possible mismatch in oxygen delivery and oxygen demand. It must be noted, that the "basic" perioperative monitoring, i.e. electrocardiogram, oxygen saturation and non-invasive or invasive blood pressure measurements is not able to accurately detect hypovolemia and ongoing organ hypoperfusion. Perioperatively, patients undergoing major abdominal surgery are prone to high risk of hemodynamic instabilities and consequently relevant changes in oxygen delivery, associated with an increase in postoperative complications and length of stay in hospital. Over the last years several studies focused on early goal directed hemodynamic therapy (GDT) with strong proof for the feasibility of such algorithms and the improvement in patient's outcome with respect to certain clinical scenarios.However, there is still a debate regarding an individualized GDT approach, based on pre-procedural defined individualized hemodynamic goals yielded by an advanced haemodynamic monitoring technology. We do have to distinguish which monitoring system, invasive to non-invasive, matches the kind of estimated risk at what time best.

ELIGIBILITY:
Inclusion Criteria:

* Major abdominal procedures
* Estimated duration ≥120 minutes
* High transfusion probability
* Anticipated blood loss ≥1000 ml

Exclusion Criteria:

* Patients less than 18 years old
* ASA I or IV classification
* Heart rhythm disorders
* Advanced peripheral artery occlusive disease
* Arteriovenous shunts concerning upper extremities
* Laparoscopic abdominal procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2014-03; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Postoperative complications | 28 days

SECONDARY OUTCOMES:
Length of hospital stay (LOS) | 28 days

CONTACTS AND LOCATIONS:
Locations (1):
- Ole Broch, Kiel, Schleswig-Holstein, Germany

REFERENCES:
- [Background] Challand C, Struthers R, Sneyd JR, Erasmus PD, Mellor N, Hosie KB, Minto G. Randomized controlled trial of intraoperative goal-directed fluid therapy in aerobically fit and unfit patients having major colorectal surgery. Br J Anaesth. 2012 Jan;108(1):53-62. doi: 10.1093/bja/aer273. Epub 2011 Aug 26. PMID 21873370
- [Background] Toyama S, Shimoyama M. Goal-directed fluid therapy in patients undergoing colorectal surgery. Br J Anaesth. 2012 May;108(5):877-8; author reply 878-9. doi: 10.1093/bja/aes110. No abstract available. PMID 22499750
- [Background] Zheng H, Guo H, Ye JR, Chen L, Ma HP. Goal-directed fluid therapy in gastrointestinal surgery in older coronary heart disease patients: randomized trial. World J Surg. 2013 Dec;37(12):2820-9. doi: 10.1007/s00268-013-2203-6. PMID 24048581
- [Background] Yates DR, Davies SJ, Milner HE, Wilson RJ. Crystalloid or colloid for goal-directed fluid therapy in colorectal surgery. Br J Anaesth. 2014 Feb;112(2):281-9. doi: 10.1093/bja/aet307. Epub 2013 Sep 20. PMID 24056586
- [Background] Bennett-Guerrero E. Hemodynamic goal-directed therapy in high-risk surgical patients. JAMA. 2014 Jun 4;311(21):2177-8. doi: 10.1001/jama.2014.5306. No abstract available. PMID 24841970
- [Background] Srinivasa S, Taylor MH, Singh PP, Lemanu DP, MacCormick AD, Hill AG. Goal-directed fluid therapy in major elective rectal surgery. Int J Surg. 2014 Dec;12(12):1467-72. doi: 10.1016/j.ijsu.2014.11.010. Epub 2014 Nov 15. PMID 25463768
- [Background] Gomez-Izquierdo JC, Feldman LS, Carli F, Baldini G. Meta-analysis of the effect of goal-directed therapy on bowel function after abdominal surgery. Br J Surg. 2015 May;102(6):577-89. doi: 10.1002/bjs.9747. Epub 2015 Mar 11. PMID 25759947
- [Background] Cannesson M, Ramsingh D, Rinehart J, Demirjian A, Vu T, Vakharia S, Imagawa D, Yu Z, Greenfield S, Kain Z. Perioperative goal-directed therapy and postoperative outcomes in patients undergoing high-risk abdominal surgery: a historical-prospective, comparative effectiveness study. Crit Care. 2015 Jun 19;19(1):261. doi: 10.1186/s13054-015-0945-2. PMID 26088649
- [Background] Hunsicker O, Scott MJ, Miller TE, Baldini G, Feldheiser A. Gastrointestinal morbidity as primary outcome measure in studies comparing crystalloid and colloid within a goal-directed therapy. Br J Anaesth. 2015 Jul;115(1):128-9. doi: 10.1093/bja/aev181. No abstract available. PMID 26089448
- [Background] Gottlieb M, Bailitz J. Comparison of Early Goal-Directed Therapy With Usual Care for Severe Sepsis and Septic Shock. Ann Emerg Med. 2015 Dec;66(6):632-4. doi: 10.1016/j.annemergmed.2015.05.025. Epub 2015 Jun 24. No abstract available. PMID 26116223
- [Background] Correa-Gallego C, Tan KS, Arslan-Carlon V, Gonen M, Denis SC, Langdon-Embry L, Grant F, Kingham TP, DeMatteo RP, Allen PJ, D'Angelica MI, Jarnagin WR, Fischer M. Goal-Directed Fluid Therapy Using Stroke Volume Variation for Resuscitation after Low Central Venous Pressure-Assisted Liver Resection: A Randomized Clinical Trial. J Am Coll Surg. 2015 Aug;221(2):591-601. doi: 10.1016/j.jamcollsurg.2015.03.050. Epub 2015 Apr 7. PMID 26206652